CLINICAL TRIAL: NCT05544201
Title: Gamma-band High-definition Transcranial Alternating Current Stimulation (HD-tACS) for Sleep Disturbances in Mild Neurocognitive Disorders Due to Alzheimer's Disease
Brief Title: Transcranial Alternating Current Stimulation (TACS) for Sleep Disturbances in Neurocognitive Disorders Due to Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, LU Hanna, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: RGC14111021
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Brain Stimulation; Alzheimer Disease; tACS; Sleep Disturbance; Aging; Cognitive Impairment, Mild
MeSH Terms: conditions — Alzheimer Disease; Parasomnias; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 40 Hz HD-tACS (Experimental): The stimulation parameters of HD-tACS include: 20 minutes at 40 Hz, 2 milliamps.
  Interventions: Device: High-definition transcranial current stimulation
- HD-tDCS (Active Comparator): The stimulation parameters of HD-tDCS include: 20 minutes at 2 milliamps, 20 seconds fade-in and 20 seconds fade-out.
  Interventions: Device: High-definition transcranial current stimulation
- Sham HD-tCS (Sham Comparator): In sham condition, the stimulation only last for 30 seconds with the electrodes left in place for a further 20 minutes. This procedure mimics the transient skin sensation of tingling induced by active HD-tACS and HD-tDCS without producing any sustainable effects.
  Interventions: Device: High-definition transcranial current stimulation

INTERVENTIONS:
Device: High-definition transcranial current stimulation — High-definition transcranial current stimulation (HD-tCS) is delivered by a battery driven direct current stimulator (DC-Stimulator Plus, NeuroConn, Ilmenau, Germany) through a central anodal electrode surrounded by four return cathodal electrodes.

SUMMARY:
Background: Sleep disturbances are highly prevalent in ageing population and patients with age-related neurodegenerative diseases, which severely affect cognition and even lead to accumulated amyloid-β (Aβ). At present, non-pharmacological interventions for sleep disturbances in dementia patients are accepted as first line of treatment, of which the evidence from clinical trials is very limited. Encouraging results from recent studies on transcranial direct current stimulation (tDCS) showed moderate positive effects on sleep quality in preclinical Alzheimer's disease (AD). Compared to tDCS, high-definition transcranial alternating current stimulation (HD-tACS) enables the entrainment of neuronal activities with optimized focality through injecting small electric current with a specific frequency and has significant enhancement effects on slow wave activities.

Objectives: The investigators aim to 1) investigate and compare the safety, efficacy and sustainability of 40 Hz HD-tACS and HD-tDCS over left dorsolateral prefrontal cortex (DLPFC) in mild neurocognitive disorder due to AD (NCD-AD) patients with sleep disturbances; 2) examine the relationship between the changes in sleep quality, cognitive function and saliva Aβ levels.

Methods: Chinese right-handed mild NCD-AD patients with sleep disturbances (aged from 60 to 90 years) will be randomly assigned to a 4-week intervention of either HD-tACS, HD-tDCS, or sham HD-tCS, with 33 participants per arm. Before intervention, structural magnetic resonance imaging (MRI) data is used to construct individual realistic head model. Comprehensive assessments, including sleep quality, cognitive performance and saliva Aβ levels will be conducted at baseline, 4th week, 8th week, 12th week and 24th week. Program adherence and adverse effects will be monitored throughout intervention.

Data analysis: The primary outcomes will be the changes in sleep quality and memory performance with modality-driven paradigms (HD-tACS, HD-tDCS, sham HD-tCS), and comparisons of group differences across different time points. Secondary outcomes will be the changes objective sleep pattern, global cognition, saliva Aβ levels and quality of life. Intention-to-treat analysis will be carried out. Changes of efficacy indicators from baseline to each follow up point will be tested with mixed effect model.

Significance: This study aims to investigate the feasibility, safety and efficacy of HD-tACS and HD-tDCS over left DLPFC for sleep disturbances and cognitive dysfunction in mild NCD-AD patients. It wills also test the program adherence, tolerability and adverse effects of this innovative neurotechonology. Information will be helpful for in-depth understanding the relationship of "sleep disturbances-amyloid deposition" and guiding the further studies of sleep medicine and neurodegenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

* Chinese, aged from 60 to 90 years.
* Mild neurocognitive disorder due to Alzheimer's disease (NCD-AD) is diagnosed according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5). NCD-AD patients are deﬁned by the following criteria: (1) evidence of modest cognitive decline in at least one of six domains of cognition (memory, perceptual- motor, complex attention, language, executive function and social cognition), and with clinical features indicative of AD, identiﬁed with the Montreal Cognitive Assessment (MoCA) score range from 22 to 26; (2) no interference with independence in everyday activities; (3) and no better explanation by other psychiatric disorders. NCD-AD patients fulﬁll the criteria of NCD and have impaired episodic memory assessed by delayed recall.
* Sleep disturbances are defined as a Pittsburgh Sleep Quality Index (PSQI) total score above 5.

Exclusion Criteria:

* Previous diagnosis of other major neurocognitive disorders;
* Past history of bipolar disorders or psychosis;
* Physically frail affecting attendance to training sessions;
* Already attending regular training, such as cognitive behavioral therapy;
* Taking a psychotropic or other medication known to affect cognition (e.g. anti-dementia medication);
* Significant communicative impairments.
* History of major neurological deficit including stroke, transient ischemic attack or brain tumor.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Pittsburg Sleep Quality Index (PSQI) | 24 weeks
  The PSQI is a 19-item questionnaire that includes seven areas of subjective sleep quality and patterns in adults over the last month including the following components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, SDs, use of sleeping medications, and daytime dysfunction (Buysse et al., 1988). Each item in the scale is scored from 0 to 3 scale (0 = no difficulty; 3 = severe difficulty). The scores are added to yield a global score ranging from 0 to 21 (0 = no difficulty; 21 = severe difficulties in all areas). This scale has good reliability and validity psychometrics and is widely used in research: Cronbach's alpha (0.77 to 0.83), sensitivity (89.6%), specificity (86.5%)(Buysse et al., 1988). Greater score of PSQI indicates worse sleep quality.
Delayed recall of words | 24 weeks
  Word-list learning test (WLLT), consisting of sixteen semantically non-associated words, is presented consecutively over three free trials of immediate recall, a 20-min delayed recall (to prevent recency effects) (Lu et al., 2018). The raw numbers of words recalled are used to assess the memory function.

SECONDARY OUTCOMES:
Efficacy evaluated by attention function performance | 24 weeks
  Attention network function measured by computerized attention network test (ANT)
Efficacy evaluated by executive function performance | 24 weeks
  Executive function is measured by category verbal fluency test (CVFT).
Efficacy evaluated by saliva Aβ40 and Aβ42 levels | 24 weeks
  The levels of Aβ40 and Aβ42 in the saliva samples will be quantified by enzyme-linked immunosorbent assay (ELISA)-type assays (Aurin Biotech, Inc.).

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lu H, Li J, Yang NS, Lam LCW, Ma SL, Wing YK, Zhang L. Using gamma-band transcranial alternating current stimulation (tACS) to improve sleep quality and cognition in patients with mild neurocognitive disorders due to Alzheimer's disease: A study protocol for a randomized controlled trial. PLoS One. 2023 Aug 4;18(8):e0289591. doi: 10.1371/journal.pone.0289591. eCollection 2023. PMID 37540692